CLINICAL TRIAL: NCT03377699
Title: A Trial Comparing the Effect and Safety of Insulin Degludec Versus Insulin Detemir, Both in Combination With Insulin Aspart, in the Treatment of Pregnant Women With Type 1 Diabetes
Brief Title: Research Study Comparing Insulin Degludec to Insulin Detemir, Together With Insulin Aspart, in Pregnant Women With Type 1 Diabetes
Acronym: EXPECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-4300; U1111-1191-3018 (Registry Identifier: World Health organization (WHO)); 2017-000048-17 (Registry Identifier: EudraCT)
Record Dates: First submitted 2017-11-16; First posted 2017-12-19 (Actual); Results first posted 2022-04-27 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Aspart; Insulin Detemir

STUDY DESIGN:
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Insulin Degludec (Experimental): Insulin Degludec once daily and Insulin Aspart 2-4 times daily
  Interventions: Drug: Insulin degludec; Drug: Insulin Aspart
- Insulin Determir (Active Comparator): Insulin Determir once daily or twice daily and Insulin Aspart 2-4 times daily
  Interventions: Drug: Insulin Aspart; Drug: Insulin detemir

INTERVENTIONS:
Drug: Insulin degludec — Injection for subcutaneous (s.c., under the skin) use once daily. The total trial duration for subjects will be maximum 25 months
  Arms: Insulin Degludec
Drug: Insulin Aspart — Injection for subcutaneous (s.c., under the skin) use 2-4 times daily with meals. The total trial duration for subjects will be maximum 25 months
Drug: Insulin detemir — Injection for subcutaneous (s.c., under the skin) use, once daily or twice daily. The total trial duration for subjects will be maximum 25 months
  Arms: Insulin Determir

SUMMARY:
The investigators are doing this study to see the effect of insulin degludec in pregnant women with type 1 diabetes, and if it is safe to use. In this study the medicine insulin degludec is compared to another medicine called insulin detemir. Participants will either get insulin degludec or insulin detemir and take it together with a medicine called insulin aspart - which treatment participants get is decided by chance. Participants will get pre-filled insulin pens. Participants will need to take blood sugar measurements several times a day. The study will last between 10 and 25 months depending on whether participants are already pregnant when they join the study. The number of visits and the tests ( for example blood and urine samples and ultrasound scans) the participants will have also depends on whether they are pregnant at study start.

ELIGIBILITY:
Inclusion Criteria: - Female, age at least 18 years at the time of signing informed consent - Diagnosed with type 1 diabetes mellitus for at least 1 year prior to the day of screening - Treated with multiple daily subcutaneous insulin injections or continuous subcutaneous insulin infusion (CSII) or inhaled insulin for at least 90 days prior to the day of screening - The subject is planning to become pregnant within 12 months from randomisation and willing to undertake pre-pregnancy counselling or the subject is pregnant with an intrauterine singleton living foetus (gestational week 8 to 13 (+6 days)) without any observed anomalies at randomisation, confirmed by an ultrasound scan - HbA1c at screening below or equal to 8.0% (64 mmol/mol) by central laboratory Exclusion Criteria: - Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within the past 90 days prior to the day of screening - Pregnant and having proteinuria as evaluated by urine protein-to-creatinine ratio above or equal to 300 mg/g in urine sample measured at screening - Subject being treated or became pregnant with assistance of in vitro fertilisation or other medical infertility treatment - Receipt of any concomitant medication contraindicated in pregnancy according to local label within 28 days before screening and between screening and randomisation for non-pregnant subjects and 28 days before conception and between conception and randomisation for pregnant subjects - Proliferative retinopathy or maculopathy requiring acute treatment. Verified by fundus photography or pharmacologically dilated fundoscopy performed within the past 90 days prior to randomisation for non-pregnant subjects or within 28 days prior to randomisation for pregnant subjects. - History of severe hyperemesis gravidarum (requiring hospitalisation)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- Argentina (4):
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Mendoza
  - Novo Nordisk Investigational Site, Salta
- Australia (7):
  - Novo Nordisk Investigational Site, Blacktown, New South Wales
  - Novo Nordisk Investigational Site, Campbelltown, New South Wales
  - Novo Nordisk Investigational Site, St Leonards, New South Wales
  - Novo Nordisk Investigational Site, Ipswich, Queensland
  - Novo Nordisk Investigational Site, Elizabeth Vale, South Australia
  - Novo Nordisk Investigational Site, Box Hill, Victoria
  - Novo Nordisk Investigational Site, Parkville, Victoria
- Austria (3):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Innsbruck
  - Novo Nordisk Investigational Site, Vienna
- Brazil (5):
  - Novo Nordisk Investigational Site, Goiânia, Goiás
  - Novo Nordisk Investigational Site, Curitiba, Paraná
  - Novo Nordisk Investigational Site, Porto Alegre, Rio Grande do Sul
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
  - Novo Nordisk Investigational Site, Ribeirão Preto
- Canada (8):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Vancouver, British Columbia
  - Novo Nordisk Investigational Site, St. John's, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Cambridge, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, PQ, Quebec
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Denmark (2):
  - Novo Nordisk Investigational Site, Aarhus N
  - Novo Nordisk Investigational Site, København Ø
- Greece (3):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Larissa
  - Novo Nordisk Investigational Site, Nea Efkarpia - Thessaloniki
- Ireland (2):
  - Novo Nordisk Investigational Site, Dublin
  - Novo Nordisk Investigational Site, Galway
- Israel (2):
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Rehovot
- Italy (5):
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Padua
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Sant'Andrea Delle Fratte (PG)
  - Novo Nordisk Investigational Site, Torino
- Russia (8):
  - Novo Nordisk Investigational Site, Kirov
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Tomsk
  - Novo Nordisk Investigational Site, Ulyanovsk
  - Novo Nordisk Investigational Site, Yekaterinburg
  - Novo Nordisk Investigational Site, Yoshkar-Ola
- Novo Nordisk Investigational Site, Belgrade, Serbia
- Novo Nordisk Investigational Site, Barcelona, Spain
- United Kingdom (10):
  - Novo Nordisk Investigational Site, Bath
  - Novo Nordisk Investigational Site, Bradford
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, High Wycombe
  - Novo Nordisk Investigational Site, Leeds
  - Novo Nordisk Investigational Site, Middlesbrough
  - Novo Nordisk Investigational Site, Norwich
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Oxford
  - Novo Nordisk Investigational Site, Truro

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Mathiesen ER, Alibegovic AC, Corcoy R, Dunne F, Feig DS, Hod M, Jia T, Kalyanam B, Kar S, Kautzky-Willer A, Marchesini C, Rea RD, Damm P; EXPECT study group. Insulin degludec versus insulin detemir, both in combination with insulin aspart, in the treatment of pregnant women with type 1 diabetes (EXPECT): an open-label, multinational, randomised, controlled, non-inferiority trial. Lancet Diabetes Endocrinol. 2023 Feb;11(2):86-95. doi: 10.1016/S2213-8587(22)00307-2. Epub 2023 Jan 6. PMID 36623517

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 56 sites in 14 countries as follows (number of sites that screened participants/number of sites that randomised participants):Argentina (5/4); Australia (7/7); Austria (3/3); Brazil (6/6); Canada (6/5); Croatia (1/1); Denmark (2/2); Greece (3/3); Ireland (2/2); Israel (2/2); Italy (5/5); Russian Federation (8/8); Serbia (2/2) and United Kingdom (8/6).
Pre-assignment Details: Based on participant pregnancy status, either non-pregnant with the intention to become pregnant or pregnant from gestational Week (GW) 8-13 + 6 days were randomised in a 1:1 ratio to receive either Insulin Degludec (IDeg) or Insulin Detemir (IDet) in combination with Insulin Aspart (IAsp) as subcutaneous injection.
Groups:
- IDeg: Participants were to receive IDeg once daily in combination with IAsp 2-4 times daily with meals as subcutaneous injection using FlexTouch and FlexPen pen injectors respectively. After randomization, the IDeg doses were adjusted once weekly to reach the glycaemic target of 4.0 - 5.0 millimoles per liter (mmol/L). It was based on mean of 3 pre-breakfast self-measured plasma glucose (SMPG) values measured on 2 days prior to visit and on the day of the visit. If one of the SMPG values was below target of 4.0 mmol/L, the insulin dose was reduced: (less than) <3.1 mmol/L: -4 units (U) and 3.1 - 3.9 mmol/L: -2U. If the mean was: 4.0-5.0 mmol/L: no adjustment; 5.1 - 10.0 mmol/L: +2U, 10.1 - 15.0 mmol/L: +4U and (greater than) >15.0 mmol/L- +6U. On the other hand, for pregnant women, the SMPG was measured 60 minutes after main meal and the IAsp doses were optimized at investigator's discretion based on the participant's SMPG values with target value (less than or equal to) ≤7.8 mmol/L.
- IDet: Participants were to receive IDet once or twice daily in combination with IAsp 2-4 times daily with meals as subcutaneous injection using FlexPen pen injector. The dose adjustments were made with a glycaemic target of 4.0 - 5.0 mmol/L. Dose adjustments: for IDet once daily - based on mean of 3 pre-breakfast SMPG values; for IDet twice daily - morning doses - based on mean pre-main evening meal SMPG values whereas the evening doses - based on mean pre-breakfast SMPG values. If one of the pre-main evening meal SMPG values were below target of 4.0 mmol/L, the insulin dose was reduced: <3.1 mmol/L: -4U and 3.1 - 3.9 mmol/L: -2U. If the mean was: 4.0-5.0 mmol/L- no adjustment; 5.1 - 10.0 mmol/L: +2U, 10.1 - 15.0 mmol/L: +4U and >15.0 mmol/L: +6U. For pregnant, the SMPG was measured 60 minutes after main meal and the IAsp doses were optimized at investigator's discretion based on the participant's SMPG values with target value (less than or equal to) ≤7.8 mmol/L.
Period: Overall Study
Arm/Group | IDeg | IDet
Started (Full analysis set for all women (FASall)) | 111 | 114
Treated (Safety analysis set for all women (SASall)) | 110 | 112
SASpregnant (Safety analysis set for pregnant women (SASpregnant)) | 91 | 94
FASpregnant (Full analysis set for pregnant women (FASpregnant)) | 92 | 96
Completed | 89 | 89
Not Completed | 22 | 25
Not completed — Withdrawal by Subject | 2 | 9
Not completed — Lost to Follow-up | 1 | 1
Not completed — Commencement of medical infertility treatment during the course of the trial | 1 | 0
Not completed — Non-pregnant subject initiating medication contraindicated during pregnancy | 1 | 1
Not completed — Randomised non-pregnant did not become pregnant and withdrawn from trial | 11 | 8
Not completed — Randomised non-pregnant did not become pregnant and NOT withdrawn from trial | 6 | 6

BASELINE CHARACTERISTICS:
Population: FASall: included all randomised women contributed to the evaluation.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg | IDet | Total
Number analyzed (Participants) | 111 | 114 | 225
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.2 (5.20) | 31.1 (5.28) | 31.2 (5.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 114 | 225
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 14 | 38
  Not Hispanic or Latino | 87 | 100 | 187
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 106 | 108 | 214
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Last Planned Glycosylated Haemoglobin (HbA1c) Prior to Delivery
Description: Mean of the HbA1c data collected at gestational week (GW) corresponding to last planned visit prior to delivery is presented. This could be either GW 16, 20, 24, 28, 32, 36. The endpoint was evaluated based on the data from both in-trial and on-treatment observation periods. In-trial observation period started at randomization and ended at the date of trial completion, up to 24 months. The date of trial completion was the date of the final scheduled follow-up visit (delivery + 58 days). For participants who had not attended the follow-up visit, the date of trial completion was the date of the last participant-investigator contact. On-treatment observation period started at the date of first dose of trial product and ended at the date of the last day on trial product, up to 22 months.
Time Frame: From GW 16 to GW 36
Population: FASpregnant included all randomised pregnant women during the trial. Overall Number of Participants Analyzed = number of participants who contributed to the analysis. Number Analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage glycosylated hemoglobin
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 84 | 84
Percentage glycosylated hemoglobin
  in-trial | 6.30 (0.70) | 6.26 (0.73)
  on-treatment: number analyzed (Participants) | 83 | 80
  on-treatment | 6.32 (0.69) | 6.26 (0.71)
Statistical Analysis 1: Comparison: IDeg vs IDet; Primary Estimand. Imputation of missing data was done within two groups of participants defined by randomised treatment arm based on a multiple imputation approach (x1000). For each of the 1000 imputed datasets last planned HbA1c prior to delivery after GW 16 was analysed using an ANCOVA with treatment, region and the stratification factor as categorical fixed effects and a pregnancy status at randomisation-by-baseline HbA1c interaction; Test type: Non-Inferiority — Non-inferiority was considered confirmed if the upper bound of the two-sided 95% CI for mean treatment difference in HbA1c is strictly below 0.4%; p < 0.0001, ANCOVA; Mean treatment difference = -0.11, 95% CI 2-sided [-0.31 to 0.08]
Statistical Analysis 2: Comparison: IDeg vs IDet; Secondary Estimand. Imputation of missing data was done within two groups of participants defined by randomised treatment arm based on a multiple imputation approach (x1000). For each of the 1000 imputed datasets last planned HbA1c prior to delivery after GW 16 was analysed using an ANCOVA with treatment, region and the stratification factor as categorical fixed effects and a pregnancy status at randomisation-by-baseline HbA1c interaction; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.3881, ANCOVA; Mean treatment difference = -0.08, 95% CI 2-sided [-0.27 to 0.11]

2. Secondary Outcome: Number of Participants With HbA1c Below or Equal to 6.0% [42 Millimoles Per Mole (mmol/Mol)] From Last Planned HbA1c Prior to Delivery (Yes/no)
Description: Number of participants who achieved pre-defined HbA1c targets ≤ 6.0% prior to delivery after GW 16 is presented. In the reported data, 'Yes' infers number of participants who have achieved ≤ 6.0% HbA1c whereas 'No' infers number of participants who have not achieved ≤ 6.0% HbA1c. The endpoint was evaluated based on the data from in-trial observation period which started at randomization and ended at the date of trial completion, up to 24 months. The date of trial completion was the date of the final scheduled follow-up visit (delivery + 58 days). For participants who had not attended the follow-up visit, the date of trial completion was the date of the last participant-investigator contact.
Time Frame: From GW 16 to GW 36
Population: FASpregnant included all randomised pregnant women during the trial. Overall Number of Participants Analyzed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 84 | 84
Participants
  Yes | 36 | 31
  No | 48 | 53

3. Secondary Outcome: Number of Participants With HbA1c Below or Equal to 6.5% (48 mmol/Mol) From Last Planned HbA1c Prior to Delivery (Yes/no)
Description: Number of participants who achieved pre-defined HbA1c targets ≤ 6.5% prior to delivery after GW 16 is presented. In the reported data, 'Yes' infers number of participants who have achieved ≤ 6.5% HbA1c whereas 'No' infers number of participants who have not achieved ≤ 6.5% HbA1c. The endpoint was evaluated based on the data from in-trial observation period which started at randomization and ended at the date of trial completion, up to 24 months. The date of trial completion was the date of the final scheduled follow-up visit (delivery + 58 days). For participants who had not attended the follow-up visit, the date of trial completion was the date of the last participant-investigator contact.
Time Frame: From GW 16 to GW 36
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 84 | 84
Participants
  Yes | 58 | 53
  No | 26 | 31

4. Secondary Outcome: Last Planned Average Post-prandial Glucose Prior to Delivery (Average of Three Main Meals)
Description: Mean of post-prandial glucose (PPG) data collected from GW 16 to last planned visit prior to delivery is presented. This could be either GW 16, 20, 24, 28, 32, 36. Average PPG is defined as the average of the available blood glucouse (BG) measurements 90 minutes after breakfast, lunch and main evening meal respectively. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period started at randomization and ended at the date of trial completion, up to 24 months. The date of trial completion was the date of the final scheduled follow-up visit (delivery + 58 days). For participants who had not attended the follow-up visit, the date of trial completion was the date of the last participant-investigator contact.
Time Frame: From GW 16 to GW 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 75 | 72
mmol/L | 7.37 (1.35) | 6.96 (1.63)

5. Secondary Outcome: Last Planned Fasting Plasma Glucose Prior to Delivery
Description: Mean of fasting plasma glucose (FPG) data collected from GW 16 to last planned visit prior to delivery is presented. This could be either GW 16, 20, 24, 28, 32, 36. The endpoint was evaluated based on the data from in-trial observation period. The in-trial observation period started at randomization and ended at the date of trial completion, up to 24 months. The date of trial completion was the date of the final scheduled follow-up visit (delivery + 58 days). For participants who had not attended the follow-up visit, the date of trial completion was the date of the last participant-investigator contact.
Time Frame: From GW 16 to GW 36
Population: FASpregnant which included all randomised pregnant women during the trial. Overall Number of Participants Analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 82 | 83
mmol/L | 6.17 (2.05) | 6.79 (2.47)

6. Secondary Outcome: Number of Hypoglycaemic Episodes During the Pregnancy Period
Description: Number of treatment emergent hypoglycaemic episodes during the pregnancy period is presented. Hypoglycaemic episode (plasma glucose <= 3.9 mmol/L (70 milligrams per decilitre (mg/dL)) Or > 3.9 mmol/L (70 mg/dL) occurring in conjunction with hypoglycaemic symptoms) is defined as treatment emergent if the onset of the episode occurs on or after the first day of trial product administration, and no later than 7 days from the last day on trial product. The endpoint was evaluated based on the data from pregnancy period. Pregnancy period started from first day of pregnancy (date of conception corresponding to the first day in GW 2) or randomisation (whichever comes last) to the date of delivery.
Time Frame: From the first day of pregnancy (date of conception) or randomisation to delivery (maximum 23 months)
Population: SASpregnant included all randomised women exposed to at least one dose of trial product and who were pregnant during the trial.
Measure: Number; unit: Episodes
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 91 | 94
Episodes | 5431 | 5982

7. Secondary Outcome: Number of Participants Who Developed Sight-threatening Retinopathy (Defined as Proliferative Retinopathy or Maculopathy) From Pregnancy Baseline to the End of Treatment (Yes/no)
Description: Sight-threatening retinopathy is defined as proliferative retinopathy or maculopathy. Eye examination was performed by fundus photography or pharmacologically dilated fundoscopy to identify if participants have developed sight-threatening retinopathy. The number of participants who developed sight-threatening retinopathy between pregnancy baseline to the end of treatment is presented. In the reported data, 'Yes' infers number of participants who developed sight-threatening retinopathy whereas 'No' infers number of participants who have not developed sight-threatening retinopathy.
Time Frame: From pregnancy baseline (corresponding to GW 8-13) to end of treatment (28 days after delivery)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 91 | 94
Participants
  Left eye: Yes | 2 | 2
  Left eye: No | 79 | 79
  Left eye: Missing | 10 | 13
  Right eye: Yes | 2 | 2
  Right eye: No | 79 | 79
  Right eye: Missing | 10 | 13

8. Secondary Outcome: Number of Participants Who Developed Sight-threatening Retinopathy Defined as Proliferative Retinopathy or Maculopathy From Treatment Baseline to the End of Treatment (Yes/no)
Description: Sight-threatening retinopathy is defined as proliferative retinopathy or maculopathy. For pregnant women, eye examination was performed by fundus photography or pharmacologically dilated fundoscopy to identify if participants have developed sight-threatening retinopathy. The number of participants who developed sight-threatening retinopathy between treatment baseline to the end of treatment is presented. In the reported data, 'Yes' infers number of participants who developed sight-threatening retinopathy whereas 'No' infers number of participants who have not developed sight-threatening retinopathy.
Time Frame: From treatment baseline (week 0) to end of treatment (28 days after delivery)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 91 | 94
Participants
  Left eye: Yes | 2 | 2
  Left eye: No | 79 | 79
  Left eye: Missing | 10 | 13
  Right eye: Yes | 2 | 2
  Right eye: No | 79 | 79
  Right eye: Missing | 10 | 13

9. Secondary Outcome: Number of Adverse Events During Pregnancy Period
Description: Number of adverse events (AEs) during pregnancy period is reported. An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. All AEs presented are treatment-emergent AEs (TEAEs). The TEAE is defined as an event that has onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment.
Time Frame: From the first day of pregnancy (date of conception) or randomisation to delivery (maximum 23 months)
Population: as for outcome 6
Measure: Number; unit: Events
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 91 | 94
Events | 429 | 328

10. Secondary Outcome: Number of Participants With Pre-eclampsia Defined as New-onset Hypertension Occurring From Gestational Week 20 to Delivery and Simultaneous Proteinuria or Presence of Eclampsia, HELLP Syndrome, or Other Severe Organ Involvement (Yes/no)
Description: Number of participants with one or more events of pre-eclampsia during pregnancy period is reported. Pre-eclampsia was defined as new-onset hypertension (greater than or equal to) ≥ 140 millimeters of mercury (mmHg) systolic or ≥ 90 mmHg diastolic, based on at least 2 measurements taken at least 4 hours apart) occurring from GW 20 to delivery and simultaneous proteinuria (defined as ≥ 300 mg protein in a 24 hours urine sample, a protein-to-creatinine ratio of ≥ 300 mg/g in a urine sample or a urine dipstick protein of 1+) or presence of eclampsia, haemolysis, elevated liver enzymes, low platelet count (HELLP) syndrome, or other severe organ involvement. In the reported data, 'Yes' infers number of participants who had pre-eclampsia events whereas 'No' infers number of participants who have not had pre-eclampsia events.
Time Frame: From GW 20 to delivery
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 91 | 94
Participants
  Yes | 12 | 7
  No | 79 | 87

11. Secondary Outcome: Number of Participants With Different Modes of Delivery e.g. Vaginal, Operative Vaginal, Planned Caesarean Section or Unplanned Caesarean Section Delivery
Description: Number of participants who had delivered by which mode of delivery (vaginal, operative vaginal, planned caesarean section or unplanned caesarean section delivery) is presented. Planned caesarean section: decision taken > 8 hours prior to delivery. Unplanned caesarean section: decision taken ≤ 8 hours prior to delivery. In case of 'early foetal death' or if the participant did not fill the pregnancy outcome form then mode of delivery was reported as 'missing'.
Time Frame: At birth
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 91 | 94
Participants
  Spontaneous vaginal birth | 11 | 18
  Planned caesarean section | 42 | 45
  Operative vaginal birth | 8 | 9
  Non planned caesarean section | 23 | 15
  Missing | 7 | 7

12. Secondary Outcome: Change in Body Weight From Pregnancy Baseline to Last Planned Visit Prior to Delivery
Description: Change in body weight from pregnancy baseline to last planned visit prior to delivery is presented.
Time Frame: From pregnancy baseline (corresponding to gestational week 8-13) to last planned visit before delivery (last weight recording before given birth)
Population: SASpregnant included all randomised women exposed to at least one dose of trial product and who were pregnant during the trial. Overall Number of Participants Analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 85 | 84
Kilogram (Kg) | 11.97 (4.79) | 10.81 (4.55)

13. Secondary Outcome: Birth Weight for Live Birth Infants
Description: Mean birth weight for live birth infants is presented. The endpoint was evaluated based on the data from in-trial observation period which started at randomization and ended at the date of trial completion, up to 24 months. The date of trial completion was the date of the final scheduled follow-up visit (delivery + 58 days). For participants who had not attended the follow-up visit, the date of trial completion was the date of the last participant-investigator contact.
Time Frame: At birth
Population: Infants who were born to FASpregnant women are included. FASpregnant is equal to randomised women who were pregnant during the trial. Overall Number of Participants Analyzed = infants with available data.
Measure: Mean (Standard Deviation); unit: grams (g)
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 86 | 84
grams (g) | 3691.0 (628.01) | 3490.2 (629.94)

14. Secondary Outcome: Birth Weight Standard Deviation (SD) Score for Live Birth Infants
Description: Mean of birth weight SD score for live infants is presented. Birth weight SD score indicates how far an infant's score deviates from the mean of the reference population of same age and same sex born at the same gestational week as per local normal curves. The SD score of 0 indicates that the infants born weigh approximately the same, negative score indicates that the infants born weigh lesser and positive score indicates that the infants born weigh more when compared with the reference population. The endpoint was evaluated based on the data from in-trial observation period which started at randomization and ended at the date of trial completion, up to 24 months. The date of trial completion was the date of the final scheduled follow-up visit (delivery + 58 days). For participants who had not attended the follow-up visit, the date of trial completion was the date of the last participant-investigator contact.
Time Frame: At birth
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Standard Deviation score
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 66 | 59
Standard Deviation score | 1.7 (1.20) | 1.2 (1.22)

15. Secondary Outcome: Number of Live Born Infants With Birth Weight < 10th Percentile for Gestational Age and Sex (Local References) (Yes/no)
Description: Number of live born infants with birth weight <10th percentile for gestational age and sex is presented.It was assessed using local birth weight percentile curves.The unit of measure 'participants' infers number of live infants.In the reported data,'Yes' infers number of live born infants with birth weight <10th percentile for gestational age and sex whereas 'No' infers number of live born infants birth weight is not <10th percentile for gestational age and sex.Unaddressed category refers to the cases where either the parents of the infant had not given consent to share information after delivery or the participants who were withdrawn from trial and they did not give any further information or if the participants did not fill the pregnancy outcome form.Endpoint was evaluated based on the data from in-trial observation period: started at randomization and ended at the date of trial completion,up to 24 months.Date of trial completion:final scheduled follow-up visit (delivery + 58 days).
Time Frame: At birth
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 86 | 85
Participants
  Yes | 1 | 3
  No | 84 | 81
  Unaddressed | 1 | 1

16. Secondary Outcome: Number of Live Born Infants With Birth Weight > 90th Percentile for Gestational Age and Sex (Local References) [Yes/no]
Description: Number of live born infants with birth weight >90th percentile for gestational age and sex is presented.It was assessed using local birth weight percentile curves.The unit of measure 'participants' infers number of live infants. In the reported data,'Yes' infers number of live born infants with birth weight >90th percentile for gestational age and sex whereas 'No' infers number of live born infants birth weight is not >90th percentile for gestational age and sex.Unaddressed category refers to cases where either parents of the infant had not given consent to share information after delivery or the participants who were withdrawn from trial and they did not give any further information or if THE participants did not fill the pregnancy outcome form.The endpoint was evaluated based on the data from in-trial observation period:started at randomization and ended at the date of trial completion,up to 24 months. Date of trial completion:final scheduled follow-up visit (delivery + 58 days).
Time Frame: At birth
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 86 | 85
Participants
  Yes | 55 | 43
  No | 30 | 41
  Unaddressed | 1 | 1

17. Secondary Outcome: Number of Participants With Pre-term Delivery
Description: Number of pregnant women who had pre-term delivery is presented. Pre-term delivery refers to delivery in < 37 completed GWs. In the reported data, 'Yes' infers number of participants who had pre-term delivery whereas 'No' infers number of participants who has not had pre-term delivery. Unaddressed category refers to the cases where either the parents of the infant had not given consent to share information after delivery or the participants who were withdrawn from trial and they did not give any further information or if the participants did not fill the pregnancy outcome form. The endpoint was evaluated based on the data from in-trial observation period which started at randomization and ended at the date of trial completion,up to 24 months. The date of trial completion was the date of the final scheduled follow-up visit (delivery+58 days). For participants who had not attended the follow-up visit,the date of trial completion was the date of the last participant-investigator contact.
Time Frame: At birth
Population: FASpregnant included all randomised women who were pregnant during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 92 | 96
Participants
  Yes | 34 | 26
  No | 57 | 66
  Unaddressed | 1 | 4

18. Secondary Outcome: Number of Participants With Early Foetal Death (Delivery Before 20 Completed GWs) (Yes/no)
Description: Number of participants who had early foetal death (delivery before 20 completed GWs) is presented. In the reported data, 'Yes' infers early foetal deaths whereas 'No' infers no foetal deaths. Unaddressed category refers to the cases where either the parents of the infant had not given consent to share information after delivery or the participants who were withdrawn from trial and they did not give any further information or if the participants did not fill the pregnancy outcome form. The endpoint was evaluated based on the data from in-trial observation period which started at randomization and ended at the date of trial completion, up to 24 months. The date of trial completion was the date of the final scheduled follow-up visit (delivery + 58 days). For participants who had not attended the follow-up visit, the date of trial completion was the date of the last participant-investigator contact.
Time Frame: At birth
Population: FASpregnant included all randomised women who were pregnant during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 92 | 96
Participants
  Yes | 4 | 5
  No | 87 | 87
  Unaddressed | 1 | 4

19. Secondary Outcome: Number of Participants Who Had Perinatal Mortality (Death of Foetus/Infant ) (Yes/no)
Description: Number of participants who had foetal/infant loss at delivery is presented. Perinatal mortality: death of foetus/infant between ≥ 20 completed GWs before delivery and <1 completed week after delivery). In the reported data, 'Yes' infers early foetal/infant deaths whereas 'No' infers no foetal/infant deaths. Unaddressed category refers to the cases where either the parents of the infant had not given consent to share information after delivery or the participants who were withdrawn from trial and they did not give any further information or if the participants did not fill the pregnancy outcome form. The endpoint was evaluated based on the data from in-trial observation period: started at randomization and ended at the date of trial completion, up to 24 months. Date of trial completion: final scheduled follow-up visit (delivery + 58 days).
Time Frame: Between at least 20 completed GWs before delivery and before 7 completed days after delivery
Population: FASpregnant included all randomised women who were pregnant during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 92 | 96
Participants
  Yes | 0 | 0
  No | 91 | 92
  Unaddressed | 1 | 4

20. Secondary Outcome: Number of Participants Who Had Neonatal Mortality (Death of Infant) (Yes/no)
Description: Number of participants who had infant loss after delivery is presented. Neonatal mortality: death of infant between ≥7 completed days after delivery and < 28 completed days after delivery. In the reported data, 'Yes' infers infant deaths whereas 'No' infers no infant deaths. Unaddressed category refers to the cases where either the parents of the infant had not given consent to share information after delivery or the participants who were withdrawn from trial and they did not give any further information or if the participants did not fill the pregnancy outcome form. The endpoint was evaluated based on the data from in-trial observation period which started at randomization and ended at the date of trial completion, up to 24 months. The date of trial completion was the date of the final scheduled follow-up visit (delivery + 58 days). For participants who had not attended the follow-up visit, the date of trial completion was the date of the last participant-investigator contact.
Time Frame: Between at least 7 completed days after delivery and before 28 completed days after delivery
Population: FASpregnant is equal to randomised women who were pregnant during the trial. Overall Number of Participants Analyzed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 92 | 96
Participants
  Yes | 0 | 0
  No | 91 | 92
  Unaddressed | 1 | 4

21. Secondary Outcome: Number of Participants With Presence of Major Abnormalities (Classified According to European Concerted Action on Congenital Anomalies and Twins (EUROCAT)) in Their Foetus/Infants
Description: Number of participants who delivered foetuses/infants with abnormalities (classified according to EUROCAT) is presented. Presence of major abnormalities were based on adjudicated data, as after adjudication congenital anomalies were classified into major or minor anomalies or in other categories. In reported data, 'Yes' infers presence of major abnormalities whereas 'No' infers absence of major abnormalities in foetus/infant. The endpoint was evaluated based on the data from in-trial observation period: started at randomization and ended at the date of trial completion up to 24 months. Date of trial completion : final scheduled follow-up visit (delivery + 58 days).
Time Frame: At birth
Population: FASpregnant included all randomised women who were pregnant during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 92 | 96
Participants
  Yes | 8 | 8
  No | 84 | 88

22. Secondary Outcome: Number of Participants With Live Born Infants (Yes/no)
Description: Number of participants with live born infants is presented. In the reported data, 'Yes' infers number of live infants whereas 'No' infers early foetal death or termination of pregnancy (induced/elective abortion). The endpoint was evaluated based on the data from in-trial observation period which started at randomization and ended at the date of trial completion, up to 24 months. The date of trial completion was the date of the final scheduled follow-up visit (delivery + 58 days). For participants who had not attended the follow-up visit, the date of trial completion was the date of the last participant-investigator contact.
Time Frame: At birth
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 92 | 96
Participants
  Yes | 86 | 85
  No | 5 | 7
  Unaddressed | 1 | 4

23. Secondary Outcome: Number of Adverse Events in the Infant
Description: AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. AEs in foetus/infant with particular focus on the AEs from delivery to follow-up are presented.
Time Frame: From delivery to final follow-up 30 days after delivery
Population: Infants who were born to SASpregnant women are included. SASpregnant were randomised women exposed to at least one dose of trial product and who were pregnant during the trial. Overall Number of Participants Analyzed = infants with available data.
Measure: Number; unit: Events
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 91 | 94
Events | 164 | 150

24. Secondary Outcome: Neonatal Hypoglycaemic Episodes Defined as Plasma Glucose Below or Equal to 1.7 mmol/L (31 mg/dL) or Below or Equal to 2.5 mmol/L (45 mg/dl) (Yes/no)
Description: Number of infants with neonatal hypoglycaemic episodes is presented. Neonatal hypoglycaemic episodes defined as plasma glucose ≤ 1.7 mmol/L (31 mg/dL) during the first 24 hours after birth or below or equal to 2.5 mmol/L (45 mg/dl) between 24 hours and 48 hours after birth. In the reported data, 'Yes' infers number of infants with neonatal hypoglycaemic episodes whereas 'No' infers number of infants with no neonatal hypoglycaemic episodes. Unaddressed category refers to the cases where either the parents of the infant had not given consent to share information after delivery or the participants who were withdrawn from trial and they did not give any further information or if the participants did not fill the pregnancy outcome form.
Time Frame: During between 24 and 48 hours after birth
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | IDeg | IDet
Number analyzed (Participants) | 86 | 85
Participants
  During the first 24 hours after birth: Yes | 20 | 19
  During the first 24 hours after birth: No | 64 | 65
  During the first 24 hours after birth: Unaddressed category | 2 | 1
  Between 24 hours and 48 hours after birth: Yes | 4 | 5
  Between 24 hours and 48 hours after birth: No | 77 | 78
  Between 24 hours and 48 hours after birth: Unaddressed category | 5 | 2

ADVERSE EVENTS:
Time Frame: For IDeg; IDet : From first day of study drug administration until final follow-up (maximum 25 months) For IDeg infants; IDet infants:From delivery until follow-up (maximum 2 months) All adverse events are TEAEs. A TEAE is defined as event that has onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomized treatment.
Description: For IDeg; IDet: SASall included all randomised women exposed to at least one dose of trial product. For IDeg infants; IDet infants: Live infants born to SASpregnant women are included. SASpregnant is equal to randomised women exposed to at least one dose of trial product and who were pregnant during the trial. AE data is presented for both participants and infants born to SASpregnat participants during the trial. Hence the total number differs from participant flow section.
Groups:
- IDegInf: Infants born to the participants who received the following treatment were included in this arm: Participants were to receive IDeg once daily in combination with IAsp 2-4 times daily with meals as subcutaneous injection using FlexTouch and FlexPen pen injectors respectively. After randomization, the IDeg doses were adjusted once weekly to reach the glycaemic target of 4.0 - 5.0 millimoles per liter (mmol/L). It was based on mean of 3 pre-breakfast self-measured plasma glucose (SMPG) values measured on 2 days prior to visit and on the day of the visit. If one of the SMPG values was below target of 4.0 mmol/L, the insulin dose was reduced: (less than) <3.1 mmol/L: -4 units (U) and 3.1 - 3.9 mmol/L: -2U. If the mean was: 4.0-5.0 mmol/L: no adjustment; 5.1 - 10.0 mmol/L: +2U, 10.1 - 15.0 mmol/L: +4U and (greater than) >15.0 mmol/L- +6U. On the other hand, for pregnant women, the SMPG was measured 60 minutes after main meal and the IAsp doses were optimized at investigator's discretion based on the participant's SMPG values with target value (less than or equal to) ≤7.8 mmol/L.
- IDetInf: Infants born to the participants who received the following treatment were included in this arm: Participants were to receive IDet once or twice daily in combination with IAsp 2-4 times daily with meals as subcutaneous injection using FlexPen pen injector. The dose adjustments were made with a glycaemic target of 4.0 - 5.0 mmol/L. Dose adjustments: for IDet once daily - based on mean of 3 pre-breakfast SMPG values; for IDet twice daily - morning doses - based on mean pre-main evening meal SMPG values whereas the evening doses - based on mean pre-breakfast SMPG values. If one of the pre-main evening meal SMPG values were below target of 4.0 mmol/L, the insulin dose was reduced: <3.1 mmol/L: -4U and 3.1 - 3.9 mmol/L: -2U. If the mean was: 4.0-5.0 mmol/L- no adjustment; 5.1 - 10.0 mmol/L: +2U, 10.1 - 15.0 mmol/L: +4U and >15.0 mmol/L: +6U. For pregnant, the SMPG was measured 60 minutes after main meal and the IAsp doses were optimized at investigator's discretion based on the participant's SMPG values with target value (less than or equal to) ≤7.8 mmol/L.
Arm/Group | IDeg | IDet | IDegInf | IDetInf
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/112 | 4/91 | 7/94
Serious Adverse Events (participants affected / at risk) | 38/110 | 33/112 | 37/91 | 42/94
Other Adverse Events (participants affected / at risk) | 76/110 | 61/112 | 17/91 | 20/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg (N=110) | IDet (N=112) | IDegInf (N=91) | IDetInf (N=94)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood ketone body increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholestasis of pregnancy (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Diabetes mellitus management (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
Gestational oedema (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (7) | 6 (7) | 0 (0) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site hypersensitivity (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Maternal therapy to enhance foetal lung maturity (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical observation (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shortened cervix (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine contractions abnormal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine hypotonus (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ABO haemolytic disease of newborn (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital naevus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital pneumonia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital pyelocaliectasis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
External auditory canal atresia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Fracture of clavicle due to birth trauma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemangioma congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (4)
Immature respiratory system (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Kidney duplex (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimal mucocoele (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Microtia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neonatal hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 9 (9) | 1 (1)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Newborn persistent pulmonary hypertension (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Poor feeding infant (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Poor weight gain neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 9 (9) | 3 (3)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Shoulder dystocia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Systemic bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Weight decrease neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anencephaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder agenesis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteric duplication (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Foetal malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polydactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal aplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ultrasound foetal abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg (N=110) | IDet (N=112) | IDegInf (N=91) | IDetInf (N=94)
Abdominal pain (Gastrointestinal disorders) | 6 (9) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 6 (8) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 22 (22) | 16 (16) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 8 (18) | 10 (16) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 5 (6) | 7 (10) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 21 (30) | 23 (45) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 7 (10) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 8 (9) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (10) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 7 (7) | 2 (2) | 0 (0) | 0 (0)
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 5 (5) | 0 (0) | 0 (0)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 8 (8) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 6 (7) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 6 (7) | 4 (4) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 6 (6) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 11 (16) | 9 (11) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 7 (12) | 5 (5) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (8) | 6 (8) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (8)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (8) | 8 (8)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-05-31): https://cdn.clinicaltrials.gov/large-docs/99/NCT03377699/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT03377699/SAP_001.pdf